CLINICAL TRIAL: NCT04601129
Title: Advantage of a Fast-recovery Protocol for Minimally Invasive Kidney Surgery
Acronym: RREIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_21; 2019-A02271-56 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-06; First posted 2020-10-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: partial nephrectomy; complete nephrectomy; minimally invasive surgery; enhanced recovery after surgery; fast track surgery
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: undergoing a minimally invasive nephrectomy, eligible to an Enhanced Recovery After Surgery Program.
  Interventions: Procedure: enhanced recovery after surgery program

INTERVENTIONS:
Procedure: enhanced recovery after surgery program — practice of an enhanced recovery after surgery program, according to the international reviews of literature and national recommendation

SUMMARY:
Shorten the time spent in the hospital (hospitalization duration) by optimizing the pre, per and postoperative care is of major medical and economic importance.

Minimally invasive surgery allows a faster recovery than open surgery. However, we need to ensure an early and secure return to normality in order to discharge patients safely from the hospital.

Clinical and biological parameters need to be controlled post-surgery.

This work is going to evaluate the efficacity of a fast - recovery program with incoming patients receiving minimally invasive surgery (laparoscopic or robotic) of partial and total nephrectomy.

The implementation of a medical and surgical fast-recovery program could

* Lower the average duration of stay in hospital (at least by 1 day) with no increase of morbidity
* Insure the absence of complications after 6 months home

DETAILED DESCRIPTION:
Prospective study of a fast recovery program evaluating the impact on the hospitalization length and the incidence of re-hospitalization for complications for 60 patients undergoing a minimally invasive nephrectomy.

The cohort will beneficiate of an extra preoperative information about the enhanced recovery after surgery program, they will benefit from a strategie of low morphine consumption during the per end post operative phase, they should need no bladder or abdominal drainage, they're encourage to eat and drink a few hours after surgery, the intravenous fluid is interrupted as early as possible, and the patients are encourage to sit, stand up and get dressed as soon as they are capable.

A form completed by the patient registers their every day capabilities to eat, drink, move, and their limitations due to pain, dizziness, and nausea. Their bowel and urine transit are also registered. This form is complete until discharge from the hospital.

Their laboratory test is monitored to identify kidney insufficiency or anemia and compared with the preoperative laboratory tests.

The hospital discharge is allowed after medical and surgical criteria are met in both groups.

A surgical evaluation is planned a week, one month, and 6 months after surgery with laboratory exams.

1 month after the discharge, a satisfaction questionnaire is filled up by the patient, answered by telephone.

At the 6 months post operative consultation, a questionnaire about chronic pain is submitted. If the patient is eligible, a chronic pain consultation is further organized.

The result will be compared to those of a retrospective cohort (+/- 60 patients) with no enhanced recovery after surgery program.

ELIGIBILITY:
Inclusion Criteria:

* Patient score from the American Society of Anesthesiologist (ASA) I, II or III stable
* Patients undergoing minimally invasive surgery (laparoscopic or robotic) partial or total unilateral nephrectomies for tumoral < pT2 stage (7 cm) with no tumor spread of the retro-peritoneal tissue, vascular or urinary tract.
* Surgery must be performed by a laparoscopic and robotic-assisted surgeon, operator must be trained using these techniques

Exclusion Criteria:

* Patient score from the American Society of Anesthesiologist (ASA) III unstable, IV and V
* Patients with renal insufficiency defined by clearance < 60 ml/min/1,73m2 (CKD-EPI)
* Patients with high embolic risk under long-term anti-coagulation medication
* Patients with congenital hemostatic deficit or antiplatelet treatment
* Patients with long term corticosteroids treatments
* History of kidney surgery or congenital unique kidney
* History of multiple abdominal surgery creating a hostile surgical environment
* intestinal chronic disease or chronic pain syndrome
* Psychiatric disorder, cognitive impairment reducing the ability to understand the discharge instructions
* Pregnant or breast-feeding women
* Patients with no social security covers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing minimally invasive surgery partial or total unilateral nephrectomies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | at 1 month

SECONDARY OUTCOMES:
Hospital readmission rate at 1 month post surgery | at 1 month
Postoperative antalgic consumption in Enhanced recovery after surgery patients | through the hospitalization, up to 5 days post surgery and long term, average of 6 months post surgery
Preoperative and postoperative Creatinine and Clearance of creatinine Delta by the CKD-EPI formula | Baseline, at 24 hours, at 1 week and at 6 months
Average Satisfaction of hospital stay and discharge on a satisfaction numerical scale | at 1 month post surgery
  Satisfaction numerical scale from 0 to 10 : with 0 being the least satisfied possible to 0 being the most satisfied possible
Neuropathic pain by Douleur Neuropathique 4 (DN4) questionnaire. | 3 and 6 months post surgery
  The questionnaire is made of 10 binnaire questions with "yes" or "no" answers, yes standing for 1 point, no standing for 0 point. The minimum score is 0 reflecting the absence of neuropathic pain, the maximum score is 10 reflecting the most intense neuropathic pain possible. The test is positive for the diagnosis of post surgical neuropathic pain at a score of 4 and above.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France